CLINICAL TRIAL: NCT02851563
Title: A Natural History Study of Canavan Disease: MGH Site
Brief Title: A Natural History Study of Canavan Disease
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2015P002400
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Canavan Disease
MeSH Terms: conditions — Canavan Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to learn more about the natural history of Canavan disease

DETAILED DESCRIPTION:
For this study, families of subjects will fill out a Canavan Patient Survey which asks questions about disease development, symptoms and progression. Patients will be seen in Dr. Eichler's Leukodystrophy clinic for standard of care appointments. These appointments will be scheduled every 6 months.

The investigators will also collect MRI images and reports that have already been done or which will be done during participation in the study on a clinical basis.

GLOBAL UNIQUE IDENTIFIERS (GUID):

A patient Global Unique Identifier (GUID) will be used as the identifier for individuals participating in the study in NeuroBANK™. The GUID is an 11-character string that is generated using encryption technology and algorithms licensed by the NCRI from the National Institutes of Health (NIH).

The GUID is generated on a secure website that utilizes 128-bit Secure Socket Layer (SSL). Of note, this website is not linked to NeuroBANK™. The GUID is generated using an irreversible encryption algorithm - it accepts twelve identifying data elements, (e.g. last name at birth, first name at birth, gender at birth, day, month and year of birth, city and country of birth, etc.), and produces a unique random-generated character string, or GUID. No identifying information is stored in the system; it is simply used to generate the GUID. If the same information is entered again, the same GUID will be returned.

The GUID is entered into NeuroBANK™ when the patient is being created in the system. As the same patient may participate in multiple studies, NeuroBANK™ will also allow capturing a study-specific ID for the patient. For more information about NeuroBANK™ or the GUID, please go to: www.neurobank.org.

Data Management:

The NCRI Data Management Team is trained and knowledgeable regarding confidentiality and integrity of data. They will be responsible for all aspects of data procedures. Alex Sherman is the ALD Connect network strategist and member of the NEALS ALS consortium. He is the director of Strategic Development and Systems of NCRI, serves on the Executive Committee of the ALS Research Group, and is one of the leaders of the NEALS ALS Consortium.

Data Quality Checks, Logic Checks and Queries:

The Data Manager (DM) at the Neurological Clinical Research Institute (NCRI) at the Massachusetts General Hospital will conduct monthly Data Quality Checks, Logic Checks, and internal data quality audits. Data field queries will be resolved in an established workflow according to the Standard Operating Procedures (SOPs). The queries may be created either at the point of entry during the data entry process, manually by the NCRI DM, or as the result of executing monthly Logic Checks.

Study-Specific Database Backup and Maintenance:

The NCRI personnel will be responsible for the database backups that will be conducted daily. Simultaneously, a separate copy of the backup in the encrypted compressed format will be maintained and saved by the System Analysts. The backups will be saved on a separate computer partition in a password-protected compressed format and also will be burnt into DVD medium and stored in a secure location.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have a confirmed diagnosis of Canavan Disease as defined by elevated NAA levels, decreased ASPA activity, or mutations in the ASPA gene.

Exclusion Criteria:

* The PI will assess whether it is in the best interest of the patient to exclude them from the study for their own comfort and well being. In cases where the PI deems it appropriate, severely affected patients will be excluded

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects Diagnosed with Canavan Disease
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-05; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure over time | baseline, 6 months, 1 year, 18 months, 2 years

SECONDARY OUTCOMES:
Change in magnetic resonance imaging findings over time | baseline, 6 months, 1 year, 18 months, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Florian Eichler, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - NYU Langone Medical Center, New York, New York
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be stored in a computer data repository at the Massachusetts General Hospital (MGH) Neurological Clinical Research Institute (NCRI). The purpose of this data repository is to capture and store data for clinical research. The repository will combine data from multiple studies. Datasets will be shared with researchers who want to advance understanding of Neurological Disease. These datasets will not contain any personal identifiable information.